CLINICAL TRIAL: NCT06645795
Title: Effect of Physiotherapy Based on Robot Assited Gait Training on Body Composition and Functional Variables in Pediatric Patient With Neurodevelopmental Alterations: Randomized and Crossover Clinical Trial
Brief Title: Robot Asissted Training on Neurodevelopmental Alterations
Acronym: RAGTNEUDEV
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Collaborators: Instituto de Investigacion Sanitaria La Fe (Other); CEE Cruz Roja Valencia (Unknown)
Responsible Party: Principal Investigator, Anna Arnal Gómez, Assistant Professor of Physiotherapy, University of Valencia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RAGT_NEUROVELOP
Record Dates: First submitted 2024-10-04; First posted 2024-10-17 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Neurodevelopmental Disorders; Cerebral Palsy
Keywords: cerebral palsy; neurodevelopmental disorders; robot assisted gait training; physical therapy; body composition; musculoeskeletal
MeSH Terms: conditions — Neurodevelopmental Disorders; Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Randomized crossover clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- robot assisted gait training plus conventional physical therapy (Experimental): Participants will complete 8 weeks of intervention of robot assisted gait training plus conventional physical therapy.
  Interventions: Combination Product: Robot assisted gait training plus conventional physical therapy
- Conventional physical therapy (Active Comparator): Participants will complete 8 weeks of conventional therapy.
  Interventions: Other: Conventional pjysical therapy

INTERVENTIONS:
Combination Product: Robot assisted gait training plus conventional physical therapy — Participants will complete 8 weeks of intervention of robot assisted gait training with the ATLAS 2030 exoskeleton (Marsi Bionics) owned by the school which they attend to. They will have 2 weekly sessions (16 sessions in total) for 4 weeks. Each session will last up to 1 hour (depending on the child's tolerance) although a minimum of 30 minutes per session and a minimum of 12 sessions will be set in this time. The training mode will be automatic. In addition, they will continue to carry out the rest of their usual treatments.
  Arms: robot assisted gait training plus conventional physical therapy
Other: Conventional pjysical therapy — Participants will complete 8 weeks of conventional therapy, with 2 sessions per week (16 sessions total). During the conventional treatment period, participants will continue with the conventional physical therapy they have received thus far. The content of the usual care treatment does not specifically address gait training, but consists of elements addressing range of motion, tone reduction, balance, activities of daily living, etc. The conventional intervention may be different for each individual based on their needs (to represent usual care), however, participants will be advised not to change the intervention, type, and frequency during the study.
  Arms: Conventional physical therapy

SUMMARY:
The aim of this randomized crossover clinical trial is to determine the effect of robot assisted gait training combined with physiotherapy on body composition and functional variables in a pediatric population with neurodevelopmental disorders.The main questions to answer are:

* Does this treatment improve body composition parameters?
* Does the treatment help maintaining functionality and without causing discomfort or pain?

Participants will perform 2 weekly physiotherapy sessions for 8 weeks, then there will be 4 weeks of washout, afer which each patient will cross over to the other group for 8 more weeks.

DETAILED DESCRIPTION:
Pediatric population with neurodevelopmental disorders, such as cerebral palsy (CP), levels IV-V of the Gross Motor Function Classification System (GMFCS), do not walk independently due to their significant physical limitations, so their body composition may be altered, which in turn affects their functional level and may lead to the appearance of musculoskeletal complications. Robot assisted gait training (RAGT) offers a new opportunity to improve mobility of pediatric population with CP levels IV-V of GMFCS, although scientific literature is still scarce in this population.

The main aim of this study is to determine the effect of RAGT on body composition and functional variables in a pediatric population with neurodevelopmental disorders. Also to analyze changes in functional, musculoeskeletal, and stress biomarkers variables after the intervention, and to evaluate the cardiorespiratory adaptation to the RAGT.

A convenience sample of 10-12 participants will be selected, who will serve as their own control. It has been taken into account that previous studies conducted on pediatric population with CP this sample size is adequate.

At the beginning of the study, 50% of the participants will be part of the RAGT group, which will perform 2 weekly sessions of RAGT plus conventional therapy; and the other 50% will belong to the conventional physical therapy group. The study consists of phases 1 and 2 of treatment with a washout period between phases: after "phase 1" (8 weeks of therapy in one of the two groups), there will be 4 weeks of washout, after which each patient will cross over to the other group in "phase 2" (for 8 weeks).

Participants will be assessed before phase 1 (T1), after phase 1 (T2), before phase 2 (T3) and after phase 2 (T4).

ELIGIBILITY:
Inclusion Criteria:

* Pediactric population with neurodevelopmental disorders who have been diagnosed with cerebral palsy.
* With a level IV or V of the GMFCS.
* Adapted to the school environment (> 6 months).
* Unable to stand without support.
* Receiving conventional physiotherapy (> 6 months).
* Receiving a standing program (standing duration at school: at least 45 minutes/day).
* With ankle orthosis.
* Meeting the specific criteria of the exoskeleton manufacturer (ATLAS 2030 Marsibionics https://www.marsibionics.com/): Weight less than 35 kg, Hip width less than 35 cm, Distance from the center of rotation of the hip to that of the knee between 24 and 33 cm, distance from the center of rotation of the knee to that of the ankle between 23 and 32 cm, the ankle can reach close to 90º with or without an orthosis, shoe size less than 33, hip and knee flexion less than or equal to 20º (even after having previously warmed up).

Exclusion Criteria:

* Severe spinal deformity.
* Severe hip dysplasia.
* Knee and hip flexion greater than 20º.
* Children treated surgically within the 1-year period prior to the evaluation date.
* Skin inflammation and open skin lesions around the trunk or limbs.
* Uncontrolled epilepsy: active epilepsy resistant to medication.
* Pacemaker, defibrillator or osteosynthesis material carriers.

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2024-10-17 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Body composition, fat % | Before phase 1 (T1, pre intervention), after phase 1 (T2, after 8 weeks intervention), before phase 2 (T3, pre intervention) and after phase 2 (T4, after 8 weeks intervention).
  Measured by bioimpedanciometry (BIA): fat (%).
Body composition, fat in kg | Before phase 1 (T1, pre intervention), after phase 1 (T2, after 8 weeks intervention), before phase 2 (T3, pre intervention) and after phase 2 (T4, after 8 weeks intervention).
  Measured by bioimpedanciometry (BIA): fat (kg)
Body composition, lean mass (kg) | Before phase 1 (T1, pre intervention), after phase 1 (T2, after 8 weeks intervention), before phase 2 (T3, pre intervention) and after phase 2 (T4, after 8 weeks intervention).
  Measured by bioimpedanciometry (BIA): lean mass (kg), lean mass (%), total mass (%), dry lean weight (%), Body mass index, and resistance at 50 kHz measured in Ohms
Body composition, lean mass (%) | Before phase 1 (T1, pre intervention), after phase 1 (T2, after 8 weeks intervention), before phase 2 (T3, pre intervention) and after phase 2 (T4, after 8 weeks intervention).
  Measured by bioimpedanciometry (BIA): lean mass (%).
Body composition, dry lean weight | Before phase 1 (T1, pre intervention), after phase 1 (T2, after 8 weeks intervention), before phase 2 (T3, pre intervention) and after phase 2 (T4, after 8 weeks intervention).
  Measured by bioimpedanciometry (BIA): dry lean weight (%).
Bone mineral density. | Before phase 1 (T1, pre intervention), after phase 1 (T2, after 8 weeks intervention), before phase 2 (T3, pre intervention) and after phase 2 (T4, after 8 weeks intervention).
  Measured by ultrasound densitometry.

SECONDARY OUTCOMES:
Functional and musculoeskeletal assessmement, clinical data. | Before phase 1 (T1, pre intervention), after phase 1 (T2, after 8 weeks intervention), before phase 2 (T3, pre intervention) and after phase 2 (T4, after 8 weeks intervention).
  Measured by the "Cerebral Palsy Follow-Up Program" (CPUP): clinical data.
Functional and musculoeskeletal assessmement, musculoskeletal history. | Before phase 1 (T1, pre intervention), after phase 1 (T2, after 8 weeks intervention), before phase 2 (T3, pre intervention) and after phase 2 (T4, after 8 weeks intervention).
  Measured by the "Cerebral Palsy Follow-Up Program" (CPUP): musculoskeletal history (previous history of fractures, subluxation or hip dysplasia), technical aids that are currently needed, neurorehabilitation treatments that are currently received at the center.
Functional and musculoeskeletal assessmement, disability assessment | Before phase 1 (T1, pre intervention), after phase 1 (T2, after 8 weeks intervention), before phase 2 (T3, pre intervention) and after phase 2 (T4, after 8 weeks intervention).
  Measured by the "Cerebral Palsy Follow-Up Program" (CPUP): disability assessment using the Pediatric Evaluation Disability Inventory (PEDI), range of motion of lower limb joints (it will be measured with a goniometer for hip, knee and ankle), spasticity in the muscles of the lower limbs (it will be measured with the modified Asworth Scale), and also the functional capacity using the Functional Mobility Scale (FMS).
Functional and musculoeskeletal assessmement, range of motion | Before phase 1 (T1, pre intervention), after phase 1 (T2, after 8 weeks intervention), before phase 2 (T3, pre intervention) and after phase 2 (T4, after 8 weeks intervention).
  Measured by the "Cerebral Palsy Follow-Up Program" (CPUP): range of motion of lower limb joints (it will be measured with a goniometer for hip, knee and ankle), spasticity in the muscles of the lower limbs (it will be measured with the modified Asworth Scale), and also the functional capacity using the Functional Mobility Scale (FMS).
Functional and musculoeskeletal assessmement, spasticity | Before phase 1 (T1, pre intervention), after phase 1 (T2, after 8 weeks intervention), before phase 2 (T3, pre intervention) and after phase 2 (T4, after 8 weeks intervention).
  Measured by the "Cerebral Palsy Follow-Up Program" (CPUP): spasticity in the muscles of the lower limbs (it will be measured with the modified Asworth Scale), and also the functional capacity using the Functional Mobility Scale (FMS).
Functional and musculoeskeletal assessmement, functional capacity | Before phase 1 (T1, pre intervention), after phase 1 (T2, after 8 weeks intervention), before phase 2 (T3, pre intervention) and after phase 2 (T4, after 8 weeks intervention).
  Measured by the "Cerebral Palsy Follow-Up Program" (CPUP): functional capacity using the Functional Mobility Scale (FMS).
Anthropometric measurements, weight | Before phase 1 (T1, pre intervention), after phase 1 (T2, after 8 weeks intervention), before phase 2 (T3, pre intervention) and after phase 2 (T4, after 8 weeks intervention).
  Weight (kg)
Anthropometric measurements, height | Before phase 1 (T1, pre intervention), after phase 1 (T2, after 8 weeks intervention), before phase 2 (T3, pre intervention) and after phase 2 (T4, after 8 weeks intervention).
  Height (cm)
Anthropometric measurements, BMI | Before phase 1 (T1, pre intervention), after phase 1 (T2, after 8 weeks intervention), before phase 2 (T3, pre intervention) and after phase 2 (T4, after 8 weeks intervention).
  Body Mass Index (kg/m2)
Anthropometric measurements, circumferences | Before phase 1 (T1, pre intervention), after phase 1 (T2, after 8 weeks intervention), before phase 2 (T3, pre intervention) and after phase 2 (T4, after 8 weeks intervention).
  circumferences of arm, calf, waist and hip (cm)
Nutritional status | Before phase 1 (T1, pre intervention), after phase 1 (T2, after 8 weeks intervention), before phase 2 (T3, pre intervention) and after phase 2 (T4, after 8 weeks intervention).
  The nutritional status of each participant will be defined by weight-for-age percentiles, height-for-age percentiles, weight-for-height ratio, and BMI-for-age, following WHO growth charts and ASPEN standards, as in previous studies in this population.
Postural ability | Before phase 1 (T1, pre intervention), after phase 1 (T2, after 8 weeks intervention), before phase 2 (T3, pre intervention) and after phase 2 (T4, after 8 weeks intervention).
  Posture and Postural Ability Scale (PPAS) in sitting, supine and prone.
Cardio-respiratory measurement, heart rate | Before phase 1 (T1, pre intervention), after phase 1 (T2, after 8 weeks intervention), before phase 2 (T3, pre intervention) and after phase 2 (T4, after 8 weeks intervention).
  Heart rate (HR) will be measured by pulse oximetry.
Cardio-respiratory measurement, oxygen saturation | Before phase 1 (T1, pre intervention), after phase 1 (T2, after 8 weeks intervention), before phase 2 (T3, pre intervention) and after phase 2 (T4, after 8 weeks intervention).
  Oxygen saturation (SaO2) will be measured by pulse oximetry.

OTHER OUTCOMES:
Parameters of the RAGT intervention, total time | During RAGT intervention sessions (8 weeks).
  During the RAGT intervention sessions, the following will also be recorded:
  Total session time (in minutes).
Parameters of the RAGT intervention, distance. | During RAGT intervention sessions (8 weeks).
  During the RAGT intervention sessions, the following will also be recorded:
  number of steps and distance walked (in metres), walking speed (the two-minute walk test will be used), spasticity of the lower limbs before and after walking with the robot (modified Asworth scale), range of motion of the lower limb joints, recording of cardiorespiratory variables during walking with an exoskeleton (HR pre and post session, SaO2 pre and post session), respiratory rate and the Physiological Cost Index will be calculated ((Working HR - Resting HR) / Walking speed).
Parameters of the RAGT intervention, walking speed | During RAGT intervention sessions (8 weeks).
  During the RAGT intervention sessions, the following will also be recorded:
  walking speed (the two-minute walk test will be used), spasticity of the lower limbs before and after walking with the robot (modified Asworth scale), range of motion of the lower limb joints, recording of cardiorespiratory variables during walking with an exoskeleton (HR pre and post session, SaO2 pre and post session), respiratory rate and the Physiological Cost Index will be calculated ((Working HR - Resting HR) / Walking speed).
Parameters of the RAGT intervention, spasticity | During RAGT intervention sessions (8 weeks).
  During the RAGT intervention sessions, the following will also be recorded:
  spasticity of the lower limbs before and after walking with the robot (modified Asworth scale).
Parameters of the RAGT intervention, range of motion | During RAGT intervention sessions (8 weeks).
  During the RAGT intervention sessions, the following will also be recorded:
  range of motion of the lower limb joints.
Parameters of the RAGT intervention, heart rate | During RAGT intervention sessions (8 weeks).
  During the RAGT intervention sessions, the following will also be recorded: cardiorespiratory variables during walking with an exoskeleton, heart rate (HR) pre and post session.
Parameters of the RAGT intervention, SaO2 | During RAGT intervention sessions (8 weeks).
  During the RAGT intervention sessions, the following will also be recorded:
  SaO2 pre and post session
Parameters of the RAGT intervention, respiratory rate | During RAGT intervention sessions (8 weeks).
  During the RAGT intervention sessions, the following will also be recorded:
  respiratory rate (cycles/minute)
Parameters of the RAGT intervention, Physiological Cost Index | During RAGT intervention sessions (8 weeks).
  During the RAGT intervention sessions, the following will also be recorded:
  Physiological Cost Index will be calculated ((Working HR - Resting HR) / Walking speed).
Pain or discomfort | Before and after the first 5 days of treatment (week 1 of each phase)
  Objectively measured by means of a saliva sample, analyzing the levels of salivary alpha-amylase (α-amylase) activity and salivary cortisol concentration. The first sample represents the child's initial stress level before the intervention program, and the second sample represents the child's stress response to the intervention. The first 5 days of conventional treatment are repeated at the same time. (Zhao, 2015) The saliva samples will be obtained using a Salivette device and processed in the favilities of IVIRMA Global Research Alliance, IVI Foundation -La Fe Health Research Institute.

CONTACTS AND LOCATIONS:
Overall Officials: ANNA ARNAL-GOMEZ, Dr., Principal Investigator — University of Valencia
Locations (1):
- University of Valencia, Valencia, València, Spain

REFERENCES:
- [Background] Engsberg JR, Ross SA, Collins DR. Increasing ankle strength to improve gait and function in children with cerebral palsy: a pilot study. Pediatr Phys Ther. 2006 Winter;18(4):266-75. doi: 10.1097/01.pep.0000233023.33383.2b. PMID 17108800
- [Background] McCormick AM, Alazem H, Zaidi S, Barrowman NJ, Ward LM, McMillan HJ, Longmuir P, Larin M, Dalton K. A randomized, cross-over trial comparing the effect of innovative robotic gait training and functional clinical therapy in children with cerebral palsy; a protocol to test feasibility. Contemp Clin Trials. 2023 Apr;127:107086. doi: 10.1016/j.cct.2023.107086. Epub 2023 Jan 17. PMID 36669727
- [Background] Peungsuwan P, Parasin P, Siritaratiwat W, Prasertnu J, Yamauchi J. Effects of Combined Exercise Training on Functional Performance in Children With Cerebral Palsy: A Randomized-Controlled Study. Pediatr Phys Ther. 2017 Jan;29(1):39-46. doi: 10.1097/PEP.0000000000000338. PMID 27984466
- [Background] Zhao X, Chen M, Du S, Li H, Li X. Evaluation of stress and pain in young children with cerebral palsy during early developmental intervention programs: a descriptive study. Am J Phys Med Rehabil. 2015 Mar;94(3):169-75; quiz 176-9. doi: 10.1097/PHM.0000000000000252. PMID 25500686